CLINICAL TRIAL: NCT05474690
Title: A Non-inferior, Randomized Controlled Phase III Clinical Study Comparing the Efficacy of TCbHPand ECHP-THP in Neoadjuvant Treatment of Operable HER2-positive Breast Cancer
Brief Title: A Study Comparing the Efficacy of TCbHP and ECHP-THP in the Neoadjuvant Treatment of HER2-positive Breast Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The new treatment plan for HER2 positive breast cancer has entered the diagnosis and treatment guide. The treatment plan ECHP-THP in this study is not the optimal treatment plan, therefore this study was terminated.
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Director, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-BC010
Record Dates: First submitted 2022-05-17; First posted 2022-07-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
Keywords: Breast cancer; HER2; pathological complete remission
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCbHP chemotherapy regimen (Active Comparator): Docetaxel + Carboplatin + Trastuzumab + Pertuzumab
  Interventions: Drug: Docetaxel + Carboplatin + Trastuzumab + Pertuzumab
- ECHP-THP chemotherapy regimen (Experimental): (Epirubicin + Cyclophosphamide - Docetaxel) + (Trastuzumab + Pertuzumab)
  Interventions: Drug: (Epirubicin + Cyclophosphamide - Docetaxel) + (Trastuzumab + Pertuzumab)

INTERVENTIONS:
Drug: Docetaxel + Carboplatin + Trastuzumab + Pertuzumab — Subjects who met the inclusion conditions were randomly divided into TCbHP group and ECHP-THP group according to 1:1.
  Stratified at randomization by the following factors: T, N, HER2 expression (HER2 protein 3+ vs HER2 protein 2+ but FISH+), and hormone receptor status (HR positive vs HR negative).
  TCbHP regimen drug dose: docetaxel 75 mg/m2 + carboplatin (AUC=6) + trastuzumab (first loading dose 8 mg/kg, sequential maintenance dose 6 mg/kg) + pertuzumab Antibiotics (the initial loading dose of 840 mg, and the sequential maintenance dose of 420 mg), every 21 days as a cycle.
  Other Names: TCbHP regimen group
  Arms: TCbHP chemotherapy regimen
Drug: (Epirubicin + Cyclophosphamide - Docetaxel) + (Trastuzumab + Pertuzumab) — Dosage of ECHP-THP regimen: epirubicin 90mg/m2+cyclophosphamide 600mg/m2 followed by docetaxel 90mg/m2, trastuzumab (first loading dose 8 mg/kg, sequential maintenance dose 6 mg /kg) + Pertuzumab (the initial loading dose of 840 mg, and the sequential maintenance dose of 420 mg), every 21 days as a cycle.
  Other Names: ECHP-THP regimen group
  Arms: ECHP-THP chemotherapy regimen

SUMMARY:
In 2020, the incidence of breast cancer surpassed that of lung cancer for the first time, becoming the number one cancer in the world. HER2 is an important prognostic indicator and therapeutic target for breast cancer. HER2-overexpressing breast cancer accounts for about 20% to 30% of all breast cancer patients. Targeted therapy for HER2 protein is the core treatment for this type of breast cancer. At present, the neoadjuvant treatment mode of trastuzumab and pertuzumab dual-target chemotherapy has become the standard neoadjuvant treatment for high-risk HER2-positive breast cancer. For patients with early-stage high-risk or locally advanced HER2-positive breast cancer, whether standard neoadjuvant regimen without anthracycline can achieve the same therapeutic effect compared with regimen containing anthracycline is still inconclusive.Therefore, this study aimed to compare the efficacy and safety of two neoadjuvant treatment regimens, TCbHP*6 and ECHP*4-THP*4, in the neoadjuvant treatment of HER2-positive breast cancer through a randomized controlled phase 3 clinical trial.

DETAILED DESCRIPTION:
Subjects were screened according to inclusion and exclusion criteria. Subjects who met the inclusion conditions were randomly divided into TCbHP group and ECHP-THP group according to 1:1.

Stratified at randomization by the following factors: T, N, HER2 expression (HER2 protein 3+ vs HER2 protein 2+ but FISH+), and hormone receptor status (HR positive vs HR negative).

1. Drug dose of TCbHP regimen: docetaxel 75 mg/m2 + carboplatin (AUC=6) + trastuzumab (first loading dose 8 mg/kg, sequential maintenance dose 6 mg/kg) + Pascal Tocilizumab (initial loading dose of 840 mg, followed by maintenance dose of 420 mg), every 21 days as a cycle.
2. Dosage of ECHP-THP regimen: epirubicin 90mg/m2 + cyclophosphamide 600mg/m2 followed by docetaxel 90mg/m2, trastuzumab (the first loading dose of 8 mg/kg, followed by maintenance The dose is 6 mg/kg) + Pertuzumab (the initial loading dose of 840 mg, and the sequential maintenance dose of 420 mg), every 21 days as a cycle.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years ≤ age ≤ 65 years, Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1；
2. Clinical T2-T4d, or T1c with axillary LN+；
3. HER2 + invasive breast cancer confirmed by histopathology Note: HER2 expression positive refers to the tumor cells with immunohistochemical staining intensity of 3 + or confirmed positive by fluorescence in situ hybridization [fish] at least once during the pathological detection/review of primary tumor in the Department of pathology of participating research center hospital；
4. Clinically measurable lesions: measurable lesions revealed by ultrasound, molybdenum target or MR (optional) within 1 month before randomization
5. Organ and bone marrow function test within one month before chemotherapy showed no chemotherapy contraindication： Absolute value of neutrophil count ≥ 2.0×10^9 / L Hemoglobin ≥ 100g / L Platelet count ≥ 100×10^9 / L Total bilirubin < 1.5 ULN (upper limit of normal value) Creatinine < 1.5 × ULN AST/ALT < 1.5×ULN
6. Echocardiography: left ventricular ejection fraction (LVEF ≥ 55%)；
7. For women of childbearing age, serum pregnancy test was negative 14 days ；
8. Signed the informed consent form prior to patient entry；

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. supraclavicular lymph node metastasis；
3. For this disease, chemotherapy, endocrine therapy, targeted therapy, reflex therapy, etc. have been received;
4. The patient has a second primary malignancy other than adequately treated skin cancer;
5. The patient has undergone major surgical procedures not related to breast cancer within 4 weeks prior to enrollment, or the patient has not fully recovered from such surgical procedures;
6. The patient has severe heart disease or discomfort, including but not limited to the following:Diagnosed history of heart failure or systolic dysfunction (LVEF < 50%)；High-risk uncontrolled arrhythmias；Angina pectoris requiring antianginal medication；Clinically significant heart valve disease；ECG showing transmural myocardial infarction；Poorly controlled high blood pressure；
7. Because the patient has other serious and uncontrollable medical diseases, the investigator believes that chemotherapy is contraindicated;
8. Known history of allergy to the drug components of this regimen; history of immunodeficiency, including HIV positive test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | up to 24 weeks
  Percentage of Participants With Pathological Complete Response (pCR) (ypT0/is/N0M0) after 6 cycles of neoadjuvant chemotherapy

SECONDARY OUTCOMES:
Number of treatment-related adverse events assessed by CTCAE v4.0 | up to 24 weeks
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 24 weeks
  Dose adjustment rate and withdrawal rate of chemotherapy drugs in two chemotherapy regimens
ORR | up to 24 weeks
  Objective response rate.ORR assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1)
DFS | up to 60 months
  From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause
OS | up to 120 months
  From date of surgery to death from any cause，whichever came first

OTHER OUTCOMES:
gene mutation rate | up to 24 weeks
  Exploring polygenic predictive models that influence PCR for different neoadjuvant regimens

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China